CLINICAL TRIAL: NCT00036842
Title: Phase II Study Of Arsenic Trioxide In Patients With Refractory Germ Cell Malignancies
Brief Title: Arsenic Trioxide in Treating Men With Germ Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069328; SWOG-S0207
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-08

CONDITIONS: Extragonadal Germ Cell Tumor; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating men who have germ cell cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (confirmed complete and partial responses) in men with refractory testicular or extragonadal germ cell malignancies treated with arsenic trioxide.
* Determine the overall and progression-free survival of patients treated with this drug.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Assess the biomarker response rate in patients with elevated biomarkers treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive arsenic trioxide IV over 1-2 hours on days 1-5. Courses repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity. Patients who achieve a confirmed complete or partial response receive up to 3 additional courses past response.

Patients are followed every 2 months for 3 years or until disease progression.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 10-40 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed testicular or extragonadal germ cell cancer
* Refractory disease, defined by at least 1 of the following criteria:

  * Disease progression during or within 4 weeks of cisplatin-containing regimen

    * Progression is defined as the appearance of new or progression of known locally advanced or metastatic disease or a rise in tumor markers (beta-human chorionic gonadotropin (beta-HCG) or alpha fetoprotein (AFP)) by at least 50% relative to the nadir
    * When the only evidence of germ cell progression or recurrence before study entry is the appearance of a new lesion in the absence of tumor marker elevation, a biopsy is required to confirm the diagnosis
  * Disease recurrence after at least 2 chemotherapy regimens, one of which includes high-dose therapy (chemotherapy with stem cell support)
  * Disease recurrence after at least 2 chemotherapy regimens and not eligible for high-dose therapy
* At least 1 of the following:

  * Unidimensionally measurable disease

    * Soft tissue, irradiated within the past 2 months, is not considered measurable
  * Elevated beta-HCG (more than 20 mIU/mL)
  * AFP greater than 2 times upper limit of normal

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Sex:

* Male

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* WBC at least 3,000/mm^3

Hepatic:

* Bilirubin less than 2.5 times upper limit of normal (ULN)
* SGOT less than 5 times ULN
* Alkaline phosphatase less than 5 times ULN

Renal:

* Creatinine no greater than 2.5 times ULN OR
* Creatinine clearance at least 40 mL/min
* Potassium normal
* Magnesium normal
* No renal dialysis

Cardiovascular:

* No prior torsades de pointes-type ventricular arrhythmia
* No prolonged QT interval (greater than 450 msec) on ECG in presence of normal potassium and magnesium

Other:

* Fertile patients must use effective contraception
* No active serious infection not controlled by antibiotics
* No known hypersensitivity to arsenic
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II disease in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* More than 28 days since prior cytotoxic agents

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 28 days since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* More than 28 days since prior experimental agents
* No concurrent or planned drugs known to prolong the QT interval

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Study Chair — OHSU Knight Cancer Institute
Locations (94):
- United States (94):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Edward Hines, Junior Hospital), Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Western New York Urology Associates, Buffalo, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Southwest Cancer and Research Center at University Medical Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Beer TM, Tangen CM, Nichols CR, Margolin KA, Dreicer R, Stephenson WT, Quinn DI, Raghavan D, Crawford ED. Southwest Oncology Group phase II study of arsenic trioxide in patients with refractory germ cell malignancies. Cancer. 2006 Jun 15;106(12):2624-9. doi: 10.1002/cncr.21925. PMID 16688776